CLINICAL TRIAL: NCT02732717
Title: The Value of Prenatal Ultrasound in the Diagnosis and Monitoring of Complicated Twin Pregnancy and Its Correlation With Chromosomal Anomalies of Twin
Brief Title: The Value of Prenatal Ultrasound in Complicated Twin Pregnancy and Its Correlation With Chromosomal Anomalies
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRS-2015-003
Record Dates: First submitted 2016-03-16; First posted 2016-04-11 (Estimated); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Complicated Twin Pregnancy
MeSH Terms: interventions — High-Energy Shock Waves; Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- abnormal ultrasound index: twin pregnancy with abnormal ultrasound index
  Interventions: Other: ultrasound (observation)
- normal ultrasound index: twin pregnancy with normal ultrasound index
  Interventions: Other: ultrasound (observation)

INTERVENTIONS:
Other: ultrasound (observation) — Important sonographic indices are to be collected from 11-14 weeks, 16-18 weeks, 22-24 weeks, 30-32 weeks and 37-39 weeks,including crown-rump length, nuchal translucency, amniotic fluid, umbilical artery flow, middle cerebral artery flow,ductus venous flow. It is observational.
  Conditions as below are thought abnormal: discordance of crown-rump length more than 20%, discordance of nuchal translucency more than 20%, either of twin with abnormal amniotic fluid (polyhydramnios or oligoamnios), either of twin with abnormal umbilical artery flow (elevated resistance index, absent or reverse diastolic flow), either of twin with abnormal middle cerebral artery flow (more than 1.5Mom), either of twin with abnormal ductus venous flow (absent or reverse a-wave).

SUMMARY:
Recent years, women with infertility have become more and more and thus assisted reproductive technology has been applied in a broad range. And the quantities of twin pregnancies are larger and larger. However, complicated twin pregnancy subsequently increased including selective intrauterine growth restriction (sIUGR), twin growth discordance, twin transfusion syndrome (TTTS) and intrauterine fetal death (IUFD). The occurrence of complicated twin pregnancy has been the leading cause of morbidity and mortality in twin and mother. Meanwhile, twin pregnancy, especially monochorionic type has suffered from higher rate of chromosomal anomalies and structural anomalies. Therefore, it is important that more attention should be paid to the prediction, clinical evaluation and the occurrence of chromosomal anomalies and structural anomalies in complicated twin pregnancy.

So far, prenatal ultrasound has been acknowledged as the best method for prenatal diagnosis and evaluation in twin pregnancy. By means of the application of prenatal ultrasound, the detection of fetal chromosome, and secondary correlation analysis, the investigators try to build prenatal ultrasound monitoring system of twin pregnancy and provide evidences for the choice of intervention and delivery time, in order to decrease the morbidity and mortality of twin and improve perinatal short and long outcomes.

The goals of this study are as below: (1) primary goal: the prediction of complicated twin pregnancy by using prenatal ultrasound; (2) primary goal: the clinical evaluation of perinatal outcomes in twin pregnancy by using prenatal ultrasound; (3) secondary goal: the analysis of the correlation between prenatal ultrasound and fetal anomalies.

DETAILED DESCRIPTION:
The study is designed as an observational prospective cohort study. The primary outcome is complicated twin pregnancy (sIUGR, TTTS, IUFD, twin growth discordance). The main exposed factors are discordance of crown-rump length more than 20%, discordance of nuchal translucency more than 20%, either of twin with abnormal amniotic fluid (polyhydramnios or oligoamnios), either of twin with abnormal umbilical artery flow (elevated resistance index, absent or reverse diastolic flow), either of twin with abnormal middle cerebral artery flow (more than 1.5Mom), either of twin with abnormal ductus venous flow (absent or reverse a-wave). Meanwhile, some demographic data are to be collected and confounding factors are to be analyzed.

Women with twin pregnancy who are examined in the department are enrolled in this study. Ultrasound will be done in 11-13+6 weeks, 16-18 weeks, 22-24 weeks, 30-32 weeks and 37-39 weeks, and perinatal outcomes are to be collected, including the diagnosis of complicated twin pregnancy, when it happens, ultrasound indices, delivery mode, delivery time, birth weight, neonatal outcomes.

When there are indications for the detection of fetal chromosome, women are probably advised to have this examination, such as non-invasive DNA, amniocentesis, umbilical cord screening, as appropriate, and written informed consent will be achieved from every patient.

ELIGIBILITY:
Inclusion Criteria:

* women with twin pregnancy starting at 11-14 weeks of gestation.

Exclusion Criteria:

* women with triplet pregnancy;
* complicating with acute internal or surgical diseases.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: pregnant women who visit the First Affiliated Hospital of Xian Jiaotong University.
Sampling Method: Non-Probability Sample
Enrollment: 580 (Estimated)
Dates: Start 2016-04; Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
the occurrence of complicated twin pregnancy as assessed by prenatal ultrasound | up to two years
  It is referred to the occurrence of at least one situation described as below. sIUGR is defined as one fetus with birth weight<the 10th percentile for gestational age and the discordance of intertwin weight is more than 20%; twin growth discordance is defined as the discordance of intertwin weight is more than 20%; TTTS:Stage I-discordant amnionic fluid volumes described as one fetus with polyhydramnios (maximum vertical pocket≥8cm) and the other fetus with oligoamnios (maximum vertical pocket<2cm), but urine is visible in the bladder of donor twin.Stage II-criteria of stage I, but urine is not visible in donor bladder.Stage III-criteria of stage II and abnormal Doppler studies of the umbilical artery, ductus venosus or umbilical vein. Stage IV-ascites or frank hydrops in either twin. Stage V-demise of either fetus;IUFD is referred to the death of twins in the uterine.

SECONDARY OUTCOMES:
without occurrence of complicated twin pregnancy as assessed by prenatal ultrasound | up to two years
  It is referred to no occurrence of any situation described as below. sIUGR is defined as one fetus with birth weight<the 10th percentile for gestational age and the discordance of intertwin weight is more than 20%; twin growth discordance is defined as the discordance of intertwin weight is more than 20%; TTTS:Stage I-discordant amnionic fluid volumes described as one fetus with polyhydramnios (maximum vertical pocket≥8cm) and the other fetus with oligoamnios (maximum vertical pocket<2cm), but urine is visible in the bladder of donor twin.Stage II-criteria of stage I, but urine is not visible in donor bladder.Stage III-criteria of stage II and abnormal Doppler studies of the umbilical artery, ductus venosus or umbilical vein. Stage IV-ascites or frank hydrops in either twin. Stage V-demise of either fetus;IUFD is referred to the death of twins in the uterine.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Han, Phd, Study Chair — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First affiliated hospital of Xian jiaotong university, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No